CLINICAL TRIAL: NCT02120274
Title: Randomized Clinical Trial to Assess the Effectiveness of Vitamin D and Vitamin B12 Supplementation in Combination With Pegylated Interferon-Alfa Plus Ribavirin for Treating Chronic Hepatitis C.
Brief Title: Vitamin D and Vitamin B12 Supplementation With Pegylated Interferon-Alfa Plus Ribavirin for Treating Chronic Hepatitis C
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: New Brazilian Guidelines for Viral Hepatitis C and Coinfetions. It does not include the treatment of chronic HCV Metavir < F3 and abandon the use of interferon.
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Henrique Pott Junior, Dr. Henrique Pott-Junior, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DB12SHCV; U1111-1155-6986 (Other: Universal Trial Number)
Record Dates: First submitted 2014-04-18; First posted 2014-04-22 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: RNA Virus Infections; Flaviviridae Infections; Hepatitis C; Hepatitis C, Chronic
Keywords: RNA Virus Infections; Flaviviridae Infections; Hepatitis C; Hepatitis C, Chronic; Vitamin D; Cholecalciferol; Vitamin B 12
MeSH Terms: conditions — RNA Virus Infections; Flaviviridae Infections; Hepatitis C; Hepatitis C, Chronic | interventions — Vitamin D; Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Pegylated Interferon-Alfa plus ribavirin for 48 weeks
- Vitamins (Experimental): Pegylated Interferon-Alfa plus ribavirin for 48 weeks together oral vitamin D 2,000 IU qd throughout, irrespective of baseline vitamin D level. Intramuscular vitamin B12 5000 UI will be given weekly in the first 12 weeks followed by a monthly injection until the end of therapy.
  Interventions: Drug: Vitamin D; Drug: Vitamin B 12

INTERVENTIONS:
Drug: Vitamin D — Oral vitamin D 2,000 IU qd throughout, irrespective of baseline vitamin D level.
  Arms: Vitamins
Drug: Vitamin B 12 — Intramuscular vitamin B12 5000 UI will be given weekly in the first 12 weeks followed by a monthly injection until the end of therapy.
  Arms: Vitamins

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the supplementation of vitamins D and B12 in combination with Pegylated Interferon-Alfa and Ribavirin in the treatment of genotype 1 chronic hepatitis C, who do not qualify to receive protease inhibitor in Brazil.

DETAILED DESCRIPTION:
Randomized clinical trial comparing rates of RVR, eRVR, EOT and SVR during standard treatment with Pegylated Interferon-Alfa plus Ribavirin compared to the same treatment supplemented with B12 and vitamin D during the treatment period.

Patients assigned to the vitamin supplementation group will receive the standard treatment of Pegylated Interferon-Alfa plus Ribavirin for 48 weeks together oral Vitamin D and intramuscular Vitamin B12. The control group will receive the same regimen of peguilated alfainterferon plus ribavirin for 48 weeks without any vitamin supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Genotype 1 HCV infection confirmed a positive test for anti-HCV antibody and detectable serum HCV RNA by PCR
* Pegylated Interferon-Alfa treatment naïve
* Liver biopsy with Metavir F2 or less
* Cognitive capacity to understand and sign the informed consent

Exclusion Criteria:

* HBV or HIV co-infection
* Hemoglobin level less than 10 g/dL or total neutrophil count less than 1,500/mm3 or platlet count below 75,000/mm3
* Creatinin ≥ 1.5 mg/dL
* Severe cardiopathy
* Pregnancy or impossibility to use birth control methods by the couple, or breast-feeding
* Conditions that, according to the investigator's judgement, preclude participation in the study, including clinical, cognitive or behavioural conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
SVR12 | 12 weeks after treatment completion
  Proportion of patients with SVR, defined as HCV RNA bellow the limit of detection 12 weeks after treatment completion with peguilated alfainterferon-2B plus ribavirin, with or without vitamin supplementation.

SECONDARY OUTCOMES:
RVR, EVR, EOT | week 4, week 12 and at the end-of-treatment.
  Proportion of patients presenting HCV RNA bellow the limit of detection at week 4 (RVR), week 12 (EVR - early virological response) and at the end-of-treatment (EOT);

CONTACTS AND LOCATIONS:
Overall Officials: Adauto Castelo, PhD, Study Director — Federal University of São Paulo; Jorge F Senise, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Outpatient Clinic of Viral Hepatitis (NUPAIG), São Paulo, São Paulo, Brazil